CLINICAL TRIAL: NCT05759871
Title: Ovarian Stimulation With FSH Alone Versus FSH Plus a GnRH Antagonist in an Oocyte Donor/Recipient Programme: a Protocol for a Non-randomised Multicenter Study
Brief Title: Ovarian Stimulation With FSH Alone Versus FSH Plus GnRH Antagonist in an Oocyte Donor/Recipient Programme
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Faculty of Medicine, School of Health Sciences, University of Thessaly, Larissa, Greece (Unknown); Embryoland, Athens, Greece (Unknown); Embryolab IVF Unit, Thessaloniki, Greece (Unknown); Assisting Nature IVF Unit, Thessaloniki, Greece (Unknown); HYGEIA IVF - Embryogenesis A.R.T. Unit, Athens, Greece (Unknown); Institute of Fertility, Athens, Greece (Unknown); Mitosis IVF Centre, Pireas, Greece (Unknown)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Professor in Obstetrics - Gynecology & Reproductive Medicine, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Non-anta-D
Record Dates: First submitted 2023-02-09; First posted 2023-03-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Premature Luteinisation; Progesterone Elevation
Keywords: Controlled ovarian stimulation; GnRH antagonist; oocyte donation; LH surge
MeSH Terms: interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-

STUDY DESIGN:
Intervention Model Description: Protocol using FSH alone with that of a protocol using FSH plus a GnRH antagonist for controlled ovarian hyperstimulation in cycles of elective freezing in the context of a donor/recipient programme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSH only (no GnRH antagonist) (Experimental): Women receive only FSH starting on day 2 of the cycle. The starting dose of FSH is 225-300 IU s.c. for the first 4 days adjusted thereafter according to the ovarian response.
  Interventions: Other: GnRH antagonist
- FSH + GnRH antagonist (Active Comparator): Women receive 225-300 IU s.c. FSH, and a GnRH antagonist from day 6 of FSH treatment at the dose of 0.25 mg per day until the triggering day. The GnRH antagonist in group 2 is injected each time immediately after the injection of FSH.
  Interventions: Other: GnRH antagonist

INTERVENTIONS:
Other: GnRH antagonist — The GnRH antagonist in the control group (standard therapy) is administered from day 6 of FSH treatment at the dose of 0.25 mg per day until the triggering day and is injected each time immediately after the injection of FSH.

SUMMARY:
The aim of this study is to compare the efficacy of a protocol using FSH alone with that of a protocol using FSH plus a GnRH antagonist for controlled ovarian hyperstimulation in cycles of elective freezing in the context of a donor/recipient programme.

DETAILED DESCRIPTION:
The hypothesis to be tested is that an ovarian stimulation protocol that includes FSH alone without any LH surge prevention regimens is not inferior to a protocol including FSH plus a GnRH antagonist in terms of clinical outcome in a donor/recipient model.

The formal sample size is calculated as follows:

If there is a true difference in favour of the experimental treatment of 5% (20% vs 15%), then 160 patients (80 per group in case of 1:1 enrolment) are required to be 80% sure that the upper limit of a one-sided 95% confidence interval (or equivalently a 90% two-sided confidence interval) will exclude a difference in favour of the standard/control group of more than 10%.

In the context of the present pilot study (as a first stage), the investigators intend to study 50 patients (25 per group in case of 1:1 enrolment). At a second stage the above mentioned sample size will be used.

ELIGIBILITY:
Inclusion Criteria:

* healthy women 21-32 years old with a BMI of 21 to 29 kg/m2 who wish to donate their oocytes
* normal ovarian reserve tests
* normal menstrual cycles of 26-32 days
* the women would not have received any hormonal treatment during the last three months before entering the study.

  * absence of coagulation and/or autoimmune disorders.

Exclusion Criteria:

1. Use of other protocols towards oocyte retrieval, such as natural, or modified natural cycles
2. Poor ovarian response according to the Bologna criteria [22],
3. History of endocrine or metabolic disorders, ovarian cystectomy or oophorectomy,
4. Women with the diagnosis of polycystic ovary syndrome
5. Clinical and/or laboratory markers of hereditary or acquired thrombophilia that complied to the standard protocols of each Unit.

   * Non-hormonal medication for a serious medical condition

Ages: 21 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Rate of LH secretory peaks | 3 weeks after start of ovarian stimulation.
  A secretory peak of LH is defined as the increase at levels ≥10 IU/l.
Rate of concentration of progesterone >1 ng/ml | At any time within 3 weeks after start of ovarian stimulation.
  Concentration of progesterone elevation >1 ng/ml

SECONDARY OUTCOMES:
Rate of ongoing clinical pregnancy | 12 weeks after last menstrual period
  Clinical pregnancy (fetal heart beat) at ultrasound
Rate of miscarriage | Within 20 weeks after last menstrual period
  Miscarriage / Loss of the embryo

OTHER OUTCOMES:
Total dose of gonadotrophins (rFSH) | 2 weeks after last menstrual period
  Dose of rFSH administered
Number of retrieved cumulus oocytes complexes (COCs) | 3 weeks after last menstrual period / and start of ovarian stimulation
  Number of retrieved cumulus oocytes complexes (COCs) at oocyte retrieval

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang HL, Lai HH, Chuang TH, Shih YW, Huang SC, Lee MJ, Chen SU. A Patient Friendly Corifollitropin Alfa Protocol without Routine Pituitary Suppression in Normal Responders. PLoS One. 2016 Apr 21;11(4):e0154123. doi: 10.1371/journal.pone.0154123. eCollection 2016. PMID 27100388
- [Background] Zhang Y, Xu Y, Yu J, Wang X, Xue Q, Shang J, Yang X, Shan X. A premature luteinizing hormone surge without elevated progesterone levels has no adverse effect on cumulative live birth rate in patient undergoing a flexible GnRH antagonist protocol: a retrospective study. J Ovarian Res. 2023 Jun 27;16(1):119. doi: 10.1186/s13048-023-01219-w. PMID 37370146
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Messinis IE, Messini CI, Anifandis G, Daponte A. Exogenous progesterone for LH surge prevention is redundant in ovarian stimulation protocols. Reprod Biomed Online. 2021 Apr;42(4):694-697. doi: 10.1016/j.rbmo.2021.01.017. Epub 2021 Jan 30. PMID 33583700
- [Background] Messinis IE, Templeton A, Baird DT. Endogenous luteinizing hormone surge in women during induction of multiple follicular development with pulsatile follicle stimulating hormone. Clin Endocrinol (Oxf). 1986 Feb;24(2):193-201. doi: 10.1111/j.1365-2265.1986.tb00762.x. PMID 3085995